CLINICAL TRIAL: NCT03801616
Title: VR 4 BR: Effects of Virtual Reality on Women Undergoing Mastectomy and Breast Reconstruction, A Pilot Study
Brief Title: Virtual Reality After Breast Reconstruction Surgery
Acronym: VR4BR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 virus
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Alice Chung, Assistant Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00055330
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Non-Opioid Pain Management; Virtual Reality
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Virtual Reality (Experimental): Every participant is provided with a VR headset
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality in controlling pain

SUMMARY:
This is a pilot study of virtual reality (VR) non-opioid management for women undergoing mastectomy and implant-based reconstruction. Study participants will receive specialized VR interventions, administered via VR headsets, to manage pain.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the effect of utilizing VR on reducing opioid use in study participants undergoing mastectomy with implant-based reconstruction compared to the control group. Investigators will follow patients throughout the course of their hospitalization and monitor outcomes including pain levels, medication requests, and satisfaction.

Eligible participants will receive a VR headset and instructed to use the VR every time they feel pain and before asking for a pain medication. They can take pain medications, if they choose to do so. At their post-op visit, study participants will be interviewed and asked questions regarding their experience with VR.

Pain level and medication use will be compared with similar individuals who undergo the same procedure but are not provided with a VR headset.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Women who plan to undergo mastectomy and implant-based reconstruction
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to read and comprehend English

Exclusion Criteria:

* Current diagnosis of epilepsy, dementia, or other neurologic disease that may prevent use of VR headset and software
* Sensitivity to flashing light
* Diagnosis of motion sickness
* Pregnancy or a medical condition where the study participant is prone to frequent nausea or dizziness
* Current or recent (less than 6 months) use of opioids
* Individuals with psychiatric disorders, including those with delirium or other disorders that may involve hallucinations or psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Implant-based reconstruction after mastectomy is not common in males.
Enrollment: 45 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chung, MD, Principal Investigator — Cedars-Sinai
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality
Started | 45
Completed | 39
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Reality
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.82051 (11.68866)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Morphine Milligram Equivalents
Description: Opioid usage is defined as mean total milligrams of morphine equivalent (MME), calculated by first multiplying the quantity of each prescribed medication by the strength of that medication (milligrams of given opioid per unit dispensed), and then multiplying this quantity-strength product by conversion factors derived from published sources to estimate the milligrams of morphine equivalent to the opioids dispensed in the prescription.
Time Frame: During hospitalization until discharge, approximately 2 days
Population: Study suspended for COVID-19 and did not re-start; terminated before the outcome measure data were collected
Arm/Group | Virtual Reality
Number analyzed (Participants) | 0

2. Secondary Outcome: Mean Difference in Pain
Description: Pain collected via ecological momentary assessment by hospital staff. Study participants will be asked by their assigned nurse to rate their pain using a standard 11-point numeric rating scale (NRS), where 0 is "no pain" and 10 is "worst imaginable pain."
Time Frame: From operation to discharge, approximately 2 days
Population: Study suspended for COVID-19 and did not re-start; terminated before the outcome measure data were collected
Arm/Group | Virtual Reality
Number analyzed (Participants) | 0

3. Secondary Outcome: Mean Difference in Length of Stay
Description: Length of stay will be collected via hospital records
Time Frame: During hospitalization until discharge, approximately 2 days
Population: Study suspended for COVID-19 and did not re-start; terminated before the outcome measure data were collected
Arm/Group | Virtual Reality
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: NA - Adverse Events not collected for this study.
Description: Study suspended for COVID-19 and did not re-start; no funding available to analyze the data
Arm/Group | Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT03801616/Prot_SAP_000.pdf